CLINICAL TRIAL: NCT00117988
Title: A Phase II Study of 17-AAG in Patients With Relapsed/Refractory CD30+ Anaplastic Large Cell Lymphoma (ALCL), Relapsed/Refractory Mantle Cell Lymphoma (MCL), and Relapsed/Refractory Classical Hodgkin's Lymphoma (HL)
Brief Title: 17-AAG in Treating Patients With Relapsed or Refractory Anaplastic Large Cell Lymphoma, Mantle Cell Lymphoma, or Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00101; NCI-2009-00101 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000433593; 2004-0792 (Other: M D Anderson Cancer Center); 6936 (Other: CTEP); P30CA016672 (NIH); R21CA117070 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2011-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2013-02

CONDITIONS: Anaplastic Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Hodgkin Disease; Lymphoma, Mantle-Cell | interventions — tanespimycin

ARMS (1):
- Arm I (Experimental): Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 1 hour on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing disease regression after completion of 8 courses may receive 2 additional courses of treatment beyond their maximal response. After completion of study treatment, patients are followed every 3 months until disease progression.
  Interventions: Drug: tanespimycin

INTERVENTIONS:
Drug: tanespimycin
  Other Names: 17-AAG

SUMMARY:
This phase II trial is studying how well 17-AAG works in treating patients with relapsed or refractory anaplastic large cell lymphoma, mantle cell lymphoma, or Hodgkin's lymphoma. Drugs used in chemotherapy, such as 17-AAG, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the complete and partial response rates and time to treatment failure in patients with relapsed or refractory anaplastic large cell lymphoma, mantle cell lymphoma, or classical Hodgkin's lymphoma treated with 17-N-allylamino-17-demethoxygeldanamycin (17-AAG).

SECONDARY OBJECTIVES:

I. Determine the safety of this drug in these patients. II. Determine the biologic effect of this drug on selected molecular targets in primary lymphoma cells from these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease type (anaplastic large cell lymphoma vs mantle cell lymphoma vs Hodgkin's lymphoma).

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 1 hour on days 1, 4, 8, and 11. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing disease regression after completion of 8 courses may receive 2 additional courses of treatment beyond their maximal response.

After completion of study treatment, patients are followed every 3 months until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during study treatment
* Must have normal organ and marrow function
* Not a candidate for stem cell transplantation
* ECOG 0-2 OR Karnofsky 60-100%
* Bilirubin normal
* Creatinine normal
* Histologically or cytologically confirmed relapsed or refractory mantle cell lymphoma, anaplastic large cell lymphoma (CD30-positive disease), or classical Hodgkin's lymphoma
* Recovered from prior biologic therapy or autologous stem cell transplantation
* Prior antibody therapy within the past 3 months allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* More than 4 weeks since prior radiotherapy (12 weeks for radioimmunotherapy) and recovered
* Recovered from prior investigational drugs
* Recovered from prior surgery
* More than 4 weeks since other prior anticancer therapy
* Concurrent low-molecular weight heparin is allowed
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm
* Absolute neutrophil count >= 1,500/mm3
* Received >= 1, but =< 3, prior treatment regimens for lymphoma (salvage therapy followed immediately by stem cell transplantation is considered 1 regimen). Single-agent monoclonal antibody therapy, cytokine therapy, or involved field radiotherapy are not considered prior treatment regimens. All prior treatments and prior antibody therapy within the past 3 months are recorded.
* Platelet count >= 75,000/mm3
* AST and ALT =< 1.5 times upper limit of normal
* Understand and provide signed informed consent.

Exclusion Criteria:

* No cardiac arrhythmia or uncontrolled dysrhythmia
* No history of myocardial infarction within the past year
* No New York Heart Association class III or IV heart failure
* No other significant cardiac disease
* No paroxysmal nocturnal dyspnea
* No oxygen requirement
* No AIDS
* No history cardiac toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubcin hydrochloride, mitoxantrone, bleomycin, or carmustine)
* No pulmonary lymphoma
* No known CNS lymphoma
* QTc >/= 450 msec for men
* QTc >/= 470 msec for women
* LVEF </= 40% by MUGA
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No symptomatic pulmonary disease requiring medication
* No significant pulmonary disease including chronic obstructive or restrictive pulmonary disease
* No dyspnea on or off exertion
* No history of pulmonary toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubcin hydrochloride, mitoxantrone, bleomycin, or carmustine)
* Not pregnant or nursing
* No other uncontrolled illness
* No other active* malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No prior allogeneic stem cell transplantation
* No history of allergic reaction to eggs
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior chest radiation or prior radiation that potentially included the heart in the field (e.g.,mantle).
* No concurrent medications that prolong or may prolong QTc
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* No prior cardiac symptoms >= grade 2
* No sufficiently compromised pulmonary status (i.e., DLCO =< 80%)
* No history of serious ventricular arrhythmia (e.g., ventricular tachycardia or ventricular fibrillation >= 3 beats in a row)
* No prior pulmonary symptoms >= grade 2
* HIV negative
* No active ischemic heart disease within 12 months.
* No congenital long QT syndrome.
* No left bundle branch block.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 02/08/2005 through 05/08/2009. All participant recruitment attempted at UT MD Anderson Cancer Center.
Groups:
- 17-AAG: 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) 220 mg/m^2 intravenous (IV) over 1 hour on days 1, 4, 8, and 11, repeated every 21 days
Period: Overall Study
Arm/Group | 17-AAG
Started | 22
Completed | 18
Not Completed | 4
Not completed — Death | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | 17-AAG
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 49.5 [25 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response
Description: Number of participants who experience complete response or partial response. Partial Response=>50% decrease in lympho node masses. Complete Response=>-75% decrease in lymph node masses.
Time Frame: Baseline to time to best response; Every 6 weeks
Population: Analysis was intention to treat (ITT). All participants with baseline and at least one post baseline target lesion measurement were included.
Measure: Number; unit: participants
Arm/Group | 17-AAG
Number analyzed (Participants) | 18
participants
  Complete Response | 0
  Partial Response | 2

ADVERSE EVENTS:
Time Frame: 4 years and 1 month
Arm/Group | 17-AAG
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 17-AAG (N=22)
Death (General disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 17-AAG (N=22)
Diarrhea (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Pain (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Fever (General disorders) | 6
Neuropathy (Nervous system disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Blurred Vision (Eye disorders) | 3
Hypertension (Cardiac disorders) | 3
Hypotension (Cardiac disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less